CLINICAL TRIAL: NCT06941506
Title: The Integration of SPOZ Technology to Support and Enhance the Vitality Acupunch Exercise Program for Improving the Cognitive Behavioral Impairment and Sensory Perceptual Impairment of Older Adults With Dementia
Brief Title: Using SPOZ Technology to Support and Enhance the Vitality Acupunch (VA) Exercise Program for Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20240009(1)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cognitive and Behavioral Impairment; Sensory and Perceptual Impairment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-SPOZ exercise program (Experimental): The VA-SPOZ exercise program was comprised of three parts: (1) the first part had 5 movements, including breathing regulation, alternating arm stretching, trunk movement, alternating left and right legs, and gradually started the blood circulation in a gentle way; (2) the second part had 14 movements, using five punching techniques, the left and right arms alternating in a natural parabola, and punching the acupoints to vibrate meridians. The purpose of the second part of the movement was to stimulate the 14 meridians and to promote the circulation of qi and blood throughout the body; (3) the third part had 5 movements, which were to adjust the breath, relax the muscles, stretch the body, and warm the face and lower back of the body by hand touch. Participants wore SPOZ devices on both hands to record and track the accuracy of the movements.The 40-minute program was administered three times a week for 6 months.
  Interventions: Other: VA-SPOZ exercise program
- Control (Active Comparator): Participants in the control group maintained their routine activities.
  Interventions: Other: Control

INTERVENTIONS:
Other: VA-SPOZ exercise program — The VA-SPOZ exercise program had three phases and took 40 minutes to complete. The program was performed in a seated position, and the participants wore SPOZ devices on both hands to record and track the accuracy of the movements.
  Arms: VA-SPOZ exercise program
Other: Control — Participants maintained their routine activities.
  Arms: Control

SUMMARY:
This project was aimed to examine the effects of a six-month VA exercise program incorporate the SPOZ technology in improving the cognitive behavioral impairment and sensory perceptual impairment of older adults with dementia in adult daycare centers.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted to examine the effects of a six-month VA exercise program incorporated the SPOZ technology in improving the cognitive behavioral impairment (using Montreal Cognitive Assessment and Neuropsychiatric Inventory Questionnaire) and sensory perceptual impairment (using Pain Assessment in Advanced Dementia) of older adults with dementia in adult daycare centers. Using convenience sampling, 10 adult daycare centers with 142 older adults were recruited, and then cluster-randomized by the daycare centers to an experimental or a control group. The experimental group received a 40-minute program 3 times a week for 6 months; the control group maintained their routine activities. The two groups were measured at three time points: before the intervention, and at three months and six months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as dementia by a physician, or
* screened by the SPMSQ as dementia
* age 65 and older

Exclusion Criteria:

* have severe cardiopulmonary disease
* have physical mobility impairment
* have spinal cord injury

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Cognitive status | 6 months
  measured by the Montreal Cognitive Assessment. A scale that includes seven aspects: visuospatial and executive functioning, animal naming, delayed recall (short-term memory), attention, language, abstraction, and orientation. The total score ranges between 0 and 30: a score ≥ 26 indicates no cognitive impairment, 18-25 indicates mild cognitive impairment, 10-17 represents moderate impairment, and < 10 indicates severe impairment.

SECONDARY OUTCOMES:
Behavioral and psychological symptoms of dementia (BPSD) | 6 months
  measured by the Neuropsychiatric Inventory Questionnaire. The 12 items measure 12 psychiatric behavioral symptoms: delusions, hallucinations, agitation/aggression, depression/bad mood, anxiety, euphoria/elation, apathy, vocally disruptive behaviors, irritable/changeable mood, aberrant motor behaviors, sleep/nighttime behaviors, and changes in appetite/eating behaviors. The assessment consists of three parts: (1) to determine the presence or absence of symptoms, 0 = no, 1 = yes; (2) to determine the severity of the symptoms, rating between 1 and 3, and the total score is 36 with higher scores indicate more severe symptoms; (3) to rate the degree of caregiver's distress caused by the client's symptoms on a scale of 0-5, and the total score is 60 with higher scores indicating greater distress.
Pain status | 6 months
  measured by the Pain Assessment in Advanced Dementia. A 5-item scale that includes patient's breathing pattern, uncomfortable/negative vocalization, facial expression, body language, and soothability. Scores are rated on a scale of 0-2. The total score is between 0 and 10; a higher score indicates a higher level of observed discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No